CLINICAL TRIAL: NCT00435877
Title: Procurement of Normal Bone, Dermis, Spleen, Thymus and Adipose Tissue for Establishment of Cell Cultures and Tissue Analyses
Brief Title: Procurement of Tissue Samples for Cell Cultures and Analyses
Status: Terminated | Type: Observational
Sponsor: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999907044; 07-D-N044
Record Dates: First submitted 2007-02-15; First posted 2007-02-16 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2012-11-05

CONDITIONS: Bone Regeneration; Fracture Healing; Cell Culture Techniques; Tissue Engineering; Differentiation
Keywords: Connective Tissue; Stromal Cells; Surgical Waste; In Vivo Studies; Tissue Analysis

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
This study will determine if bone marrow stromal cells can be used as a graft for regeneration of bony defects. These cells have the ability to form new bone and to support the formation of blood. Stromal cells have been identified in other tissues, such as the dermis (underside of skin), spleen, thymus and fat, but it is not known whether these cells can make bone and support blood formation as well as bone marrow stromal cells.

Patients undergoing surgery at Suburban Hospital in Bethesda, Maryland, in which some of the bone, dermis, spleen, thymus or fat tissue is removed may be eligible for this study.

For this study, a small piece of the tissue that is removed during surgery for examination by a pathologist will be used for research. Stromal cells from the specimen will be collected and grown in the laboratory. The genes and proteins in the different cell types will be compared, and the ability of stromal cells from the different tissues to make bone and to support the formation of blood will be studied.

DETAILED DESCRIPTION:
Background: It is now apparent that virtually every human post-natal tissue contains some type of stem/progenitor cell population that is responsible for tissue turnover and repair. Our previous studies have identified a subset of human bone marrow stromal cells (BMSCs) that is multi-potent and able to regenerate bone, cartilage, myelosupportive stroma and adipocytes, whereas stromal cells derived from human spleen (SpSCs) and thymus (TSCs) only form myelosupportive stroma. Recent studies suggest that human adipose-derived stromal cells (ASCs) may be similar to BMSCs, whereas stromal cells derived from human dermis (DSCs) have none of these properties (and serve as a negative control for most experiments in vitro and in vivo). How similar or dissimilar these different stromal cell populations are has yet to be determined. Molecular profiling is needed to compare these different populations and in order to elucidate the factors that control differentiation stromal cells into one cell type or another.

Objectives: Surgical waste (bone with red marrow, dermis, spleen, thymus and adipose tissues) from males and females of varying ages undergoing clinically indicated surgical procedures will be used to establish stromal cell cultures to study the molecular profile and differentiation capacity of the stromal cell populations from different tissues and to further characterize the regulation of gene expression and protein synthesis in these stem/progenitor cells.

Eligibility: Any patient who is undergoing clinically indicated surgery that entails removal of bone with red marrow, dermis, spleen, thymus and adipose tissue, and who do not have: 1) a history of metabolic bone disease, 2) any form of cancer or have been treated by chemotherapy or irradiation for cancer, and 3) have not received agents known to affect bone metabolism.

Design: Normal surgical waste (bone with red marrow, dermis, spleen, thymus and adipose) from procedures that are performed on males and females at Suburban Hospital will be placed in nutrient medium (provided by NIDCR) and sent to the NIDCR for the establishment of cell culture strains. Only the age, gender and site from which the tissue was removed will be recorded. The cell cultures from the different tissues will be used to determine their phenotypic character and differentiation properties by molecular profiling, and for studies to elucidate the regulation of gene expression and protein synthesis. Similarly, a portion of the samples obtained at Suburban Hospital will be used to generate histological sections of the normal tissues that will be used to screen newly developed antibodies and molecular probes. In some cases, RNA will be extracted from the tissues for RT-PCR analysis. These samples (cells, sections, mRNA) will also serve as normal controls for studies performed on samples obtained from patients with various diseases recruited to NIH under current NIH protocols (97-D-0055, 97-D-0145, 01-D-0184).

ELIGIBILITY:
* INCLUSION CRITERIA:

Any patient over the age of 18 years who is undergoing a clinically indicated or elective surgery that entails removal of bone with red marrow,periosteum, dermis, spleen, thymus, muscle and adipose tissue.

All patients must sign a document of informed consent indicating their understanding that the specimens collected and demographic information provided is only for research purposes.

EXCLUSION CRITERIA:

Any patient that has a history of metabolic bone disease.

Any patient that has cancer of any type, or has been treated for cancer of any type.

Any patient that has been treated with a reagent known to affect bone metabolism (bisphosphonates, steroids, vitamin D)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2007-01-29; Study Completion 2012-11-05

CONTACTS AND LOCATIONS:
Overall Officials: Pamela G Robey, Ph.D., Principal Investigator — National Institute of Dental and Craniofacial Research (NIDCR)
Locations (1):
- Suburban Hospital, Bethesda, Maryland, United States

REFERENCES:
- [Background] Bianco P, Riminucci M, Kuznetsov S, Robey PG. Multipotential cells in the bone marrow stroma: regulation in the context of organ physiology. Crit Rev Eukaryot Gene Expr. 1999;9(2):159-73. doi: 10.1615/critreveukargeneexpr.v9.i2.30. PMID 10445154
- [Background] Friedenstein AJ, Chailakhyan RK, Latsinik NV, Panasyuk AF, Keiliss-Borok IV. Stromal cells responsible for transferring the microenvironment of the hemopoietic tissues. Cloning in vitro and retransplantation in vivo. Transplantation. 1974 Apr;17(4):331-40. doi: 10.1097/00007890-197404000-00001. No abstract available. PMID 4150881
- [Background] Gronthos S, Franklin DM, Leddy HA, Robey PG, Storms RW, Gimble JM. Surface protein characterization of human adipose tissue-derived stromal cells. J Cell Physiol. 2001 Oct;189(1):54-63. doi: 10.1002/jcp.1138. PMID 11573204